CLINICAL TRIAL: NCT02672969
Title: The Evaluation of Pre-Post Smoke Evacuation Uses on Surgical Smoke and Bio-Aerosols in Operating Rooms at a University Hospital, Thailand
Brief Title: The Evaluation of Pre-Post Smoke Evacuation Uses on Surgical Smoke and Bio-Aerosols in Operating Rooms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Usavadee Asdornwised, Assoc.Prof.Dr., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 248/2558 (EC1)
Record Dates: First submitted 2016-01-21; First posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Smoke
Keywords: smoke evacuation system; surgical smoke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoke evacuation uses (Experimental): Smoke evacuation uses means using RapidVac Smoke Evacuator with electrosurgical unit during coagulation and cutting surgery. (Experimental group)
  Interventions: Device: RapidVac Smoke Evacuator
- no smoke evacuation uses (No Intervention): No smoke evacuation uses means using only the regular electrosurgical unit during coagulation and cutting surgery. (Control group)

INTERVENTIONS:
Device: RapidVac Smoke Evacuator — The intervention group, using the smoke evacuation (RapidVac Smoke Evacuator) in each OR, the data collection for the amount of surgical smoke and bio-aerosols' particles will be collected during pre-surgery and during surgery (every 30 mins).
  Before using the smoke evacuation, the amount of surgical smoke and bio-aerosols' particles in the surgical field and OR environment will be measured by AeroTraxTM Handheld Airborne Particle Counter. This record includes the amount and size of smoke and bio-aerosol particles in each area such as anesthetic area (anesthesiologist physicians and nurses area); instrument preparation area (circulating nurses area) and surgical area (surgeons and scrub nurses areas).
  Arms: Smoke evacuation uses

SUMMARY:
This study aims to evaluate the pre-post smoke evacuation uses on surgical smoke and bio-aerosols particles in operating rooms at a university hospital, Thailand.

DETAILED DESCRIPTION:
Purpose of Project

Smoke and bio-aerosols are routinely produced by surgical instruments; eg, lasers, electrosurgical units, radiofrequency devices, ultrasonic devices, power tools. Plume and bio-aerosols contain odor-causing and odorless toxic gases, vapors, dead and live cellular debris (including blood fragments), and viruses. These airborne contaminants can pose respiratory, ocular, dermatological and other health-related risks, including mutagenic and carcinogenic potential, to patients and operating room personnel. The National Institute of Occupational Safety and Health (NIOSH) and the Center for Disease Control (CDC) have also studied electrosurgical smoke at length. Therefore, the equipment of smoke evacuation in OR needs to be used. Therefore, this study aims to evaluate the pre-post smoke evacuation uses on surgical smoke and bio-aerosols particles in operating rooms at a university hospital, Thailand.

Methodology Association of periOperative Registered Nurses (AORN) guideline is used as the conceptual framework of this study including evidence based practice for smoke and bio-aerosols evacuation systems. The study design is a quasi-experimental study (manipulation and control only, without randomization) comparing the amount of surgical smoke and bio-aerosols particles pre- post smoke evacuation uses. The samples consist of 64 cases of surgical patients who receive head-neck or breast surgery and 64 cases of surgical patients who receive abdominal laparoscopic surgery. The amount of surgical smoke and bio-aerosols' particles in the surgical field and OR environment are measured by AeroTraxTM Handheld Airborne Particle Counter Model 9306.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients who receive head-neck or breast surgery or surgical patients who receive abdominal laparoscopic surgery

Exclusion Criteria:

* Emergency cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The amount of surgical smoke and bio-aerosols' particles in the Head, Neck & Breast/ Laparoscopic abdominal surgical field will be measured by AeroTraxTM Handheld Airborne Particle Counter Model 930 | Operating time, about 1- 3 hours
  Measuring the smoke particles and using data record for the amount of particles (particles/ft3)(millions) in 3 areas; anesthetic area, instrument preparation area, and surgical area for the Head, Neck & Breast surgery/Laparoscopic abdominal surgery

SECONDARY OUTCOMES:
The size of surgical smoke and bio-aerosols' particles in the Head, Neck & Breast /Laparoscopic abdominal surgical field will be measured by AeroTraxTM Handheld Airborne Particle Counter Model 930 | Surgical time 1-3 hours
  Measuring the particle size and using data record for size of particles (μm) (from 0.3 to 10 μm) in 3 areas; anesthetic area, instrument preparation area, and surgical area for the Head, Neck & Breast surgery/Laparoscopic abdominal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Usavadee Asdornwised, PhD, Principal Investigator — Faculty of Nursing, Mahidol University
Locations (1):
- Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barrett WL, Garber SM. Surgical smoke: a review of the literature. Is this just a lot of hot air? Surg Endosc. 2003 Jun;17(6):979-87. doi: 10.1007/s00464-002-8584-5. Epub 2003 Mar 19. PMID 12640543
- [Result] Sanderson C. Surgical smoke. J Perioper Pract. 2012 Apr;22(4):122-8. doi: 10.1177/175045891202200405. PMID 22567763
- [Result] Ball K. Compliance with surgical smoke evacuation guidelines: implications for practice. AORN J. 2010 Aug;92(2):142-9. doi: 10.1016/j.aorn.2010.06.002. PMID 20678603